CLINICAL TRIAL: NCT06118606
Title: Interventional Multidisciplinary Rehabilitation and Special Support; a Pilot Study of a Case Manager-led Multidisciplinary Intervention in ICU Survivors At Risk for Psychological or Physical Morbidity -IMPRESS-ICU Pilot Study
Brief Title: Pilot Study of a Multidisciplinary Intervention in ICU Survivors At Risk for Psychological or Physical Morbidity
Acronym: IMPRESS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Anna Milton, Principal investigator, Region Stockholm
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2022-03436-01
Record Dates: First submitted 2023-11-01; First posted 2023-11-07 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Post-Intensive Care Syndrome; Depressive Symptoms; Anxiety; Physical Disability; Posttraumatic Stress Symptom; Critical Care, Intensive Care
Keywords: Post-intensive care syndrome; Pilot study; Early follow-up intervention
MeSH Terms: conditions — postintensive care syndrome; Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Pilot study of the feasibility of the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Interventional arm (Experimental): Intervention arm
  Interventions: Other: Case-manager led multidisciplinary follow-up after intensive care

INTERVENTIONS:
Other: Case-manager led multidisciplinary follow-up after intensive care — Early in-hospital follow-up in survivors of intensive care with an increased risk of psychological/physical sequelae. The follow-up is led by a case-manager reassessing the patient after ICU discharge for psychological/physical rehabilitation needs. The CM will discuss patient needs with concerned specialists in a multidisciplinary team, leading to the establishment of a personal rehabilitation plan, communicated to the patient and next-of-kin. The CM will keep track of the patient during hospital stay and ensure primary care rehabilitation (if needed) is established once the patient is discharged from the hospital. The CM will contact the patient weekly to follow up on well-being and primary care activities until 12 weeks after discharge.

SUMMARY:
Pilot study of the feasibility and utility of an early, in-hospital multidisciplinary intervention in ICU survivors at risk for psychological and physical problems post-ICU stay

DETAILED DESCRIPTION:
60 adult patients at two hospitals in Region Stockholm (Karolinska University Hospital and Södersjukhuset) with an ICU stay ≥12 hours with increased risk for psychological/physical sequelae will be invited to participate.

Intervention: Early re-assessment and multidisciplinary follow-up, led by an ICU follow-up staff (Case Manager, CM). The CM will support the patient and coordinate the rehabilitation efforts from ICU discharge to primary care with a secondary, deepened assessment of symptoms in the ward, recapitulation and information about the time spent in the ICU, followed by a multidisciplinary discussion with concerned specialists and the set-up of an individual rehabilitation plan communicated to the patient and the informal caregivers. The CM will keep track of the patient during hospital stay and ensure that there is a plan for further primary care rehabilitation after hospital discharge. The CM will contact the patient weekly to follow up on wellbeing and planned primary care activities until 12 weeks. At twelve weeks, patients will be assessed with regards to psychological symptoms (HADS, PTSS-14) and physical disability (BI).

Outcome: The primary outcome is the feasibility of the intervention. Patients and informal caregivers will be invited to participate in semi-structured interviews that will deepen the knowledge about their views upon the intervention, needs and suggested measures to improve the patients' recovery. Resource utilisation will be documented by the CM and feedback collected from involved ICU staff and hospital clinicians. Secondary outcomes are patients' level of psychological and physical problems and health-related quality of life. The results from the pilot study will inform a subsequent randomized controlled trial of an early follow-up intervention.

ELIGIBILITY:
Inclusion Criteria:

- Patients admitted ≥12 hours to the ICU with an increased risk for physical or psychological sequelae (assessed with the PROGRESS-ICU/PREPICS instruments)

Exclusion Criteria:

* Dementia or other major cognitive problems
* Structural brain or spinal cord injury
* Multiple limitations of medical treatment
* Insufficient language skills (Swedish)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the intervention | Outcome measured during and after termination of data collection and end of intervention
  Evaluation of the method including resource utilization with involved ICU follow-up staff/case managers and patients and their informal caregivers.
Utility of the intervention | Outcome measured three-four months after ICU discharge
  Patient and caregiver views on the intervention's utility. Views on the intervention from hospital ward staff.

SECONDARY OUTCOMES:
Depressive symptoms post-ICU | Outcome measured three months after ICU discharge
  Assessment of patients' symptoms of depression post-intervention
Anxiety symptoms post-ICU | Outcome measured three months after ICU discharge
  Assessment of patients' symptoms of anxiety post-intervention
Symptoms of post-traumatic stress post-ICU | Outcome measured three months after ICU discharge
  Assessment of patients' symptoms of post-traumatic stress post-intervention
Physical disability post-ICU | Outcome measured three months after ICU discharge
  Assessment of physical performance post-intervention
Health-related quality of life post-ICU | Outcome measured three months after ICU discharge
  Health-related quality of life (HRQL) assessed with the RAND-36 questionnaire, scoring 0-100 where a higher score indicates greater HRQL.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Milton, Principal Investigator — Karolinska Institutet/Karolinska University Hospital
Locations (2):
- Sweden (2):
  - ICU Karolinska University Hospital, Stockholm
  - ICU Södersjukhuset, Stockholm

IPD SHARING:
Plan to Share IPD: No